CLINICAL TRIAL: NCT03859193
Title: Education Nutritional Video for Gestational Diabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HM20014445
Record Dates: First submitted 2019-02-27; First posted 2019-03-01 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): Participants will receive standard nutrition counseling
- Video (Experimental): Participants will watch an Nutritional video at their first high risk visit. Participants will also receive standard nutrition counseling
  Interventions: Behavioral: Nutritional Video

INTERVENTIONS:
Behavioral: Nutritional Video — A 10 - 15 minute video
  Arms: Video

SUMMARY:
The purpose of this research study is to find out if watching an educational video about nutrition helps participants learn about how different foods affect their blood sugar and how Gestational Diabetes affects pregnancy.

DETAILED DESCRIPTION:
* Patients diagnosed with gestational diabetes receive standard nutritional counseling at their first high risk clinic visit. All patients agreeing to participate in the study will at this visit fill out a knowledge questionnaire prior to receiving counseling.
* Patients will be randomized into standard counseling or standard counseling plus educational video using block randomization that has been integrated into the Redcap Survey. Once the Initial survey is completed the RedCap program will inform the patient whether they are randomized to Video or NO Video.
* Patients randomized to Video will watch the video will watch the video on a clinic designated computer. Patients randomized to no Video will not watch a video.
* At the next High risk clinic visit one to two weeks later all patients will fill out the same fill out the same questionnaire in addition to the The Problem Areas In Diabetes (PAID) questionaire.
* English-speaking patients will view the English version of the video, and Spanish-speaking patients will view the Spanish version of the video in either English or the dubbed Spanish version.
* A Spanish version of the patient hand-out will be provided in an amendment, prior to their use with Spanish- speaking patients.

ELIGIBILITY:
Inclusion Criteria:

* Any diagnosis of Diabetes in Pregnancy
* Received at least one session of nutritional counseling from the registered dieticians

Exclusion Criteria:

* Age < 18
* Patients without diagnosis of diabetes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women with a diagnosis of Diabetes in Pregnancy
Enrollment: 42 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
Change in nutritional knowledge | Baseline to 1 week
  Change in nutritional knowledge as measured by 10-item Gestational Diabetes Mellitus Knowledge Questionnaire, each question answered correctly is counted as one towards total score. Maximum score is 10, minimum score is 0.

SECONDARY OUTCOMES:
Problem Areas In Diabetes (PAID) questionnaire Score | 1 week
  Respondents are asked to indicate the degree to which each of the items is currently a problem for them, from 0 (not a problem) to 4 (a serious problem). This is a 20 item questionaire and calculates a score of 1-100
Patient Satisfaction with Care | 1 week
  Patient satisfaction on a scale of 1 to 5

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Koehn, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No